CLINICAL TRIAL: NCT04092218
Title: Prevalence of Parenting Style in Group of Children With Primary Dentition in Their First Dental Visit- A Cross Sectional Study
Brief Title: Prevalence of Parenting Style and Child Behavior
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Rouane Alaa El-Din Mohamed El-Mahdy, Principal investigator, Cairo University
Other Study IDs: Parenting style child behavior
Record Dates: First submitted 2019-09-14; First posted 2019-09-17 (Actual); Last update posted 2020-03-24 (Actual); Status verified 2020-03

CONDITIONS: Child Behavior; Parenting; Parent-Child Relations
Keywords: parenting style; child behavior; first dental visit; caries experience
MeSH Terms: conditions — Child Behavior | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Questionnaire — Data will be obtained through a written questionnaire to determine the type of parenting style of parents or caregivers.
  The collected data will be saved and tabulated on computer and finally statistically analysed.

SUMMARY:
Prevalence of parenting style and assessment of child behavior and caries experience in relation to parenting style during first dental visit.

DETAILED DESCRIPTION:
The success of dental visit depends on the child's behavior and cooperation which can be recognized from the child's first visit. Child's behavior can be affected by the parenting style. There are four types of parenting styles: authoritative, authoritarian, permissive and neglecting, each affects the child in different ways.

Recently parenting styles became very interesting since parents are the primary caregivers and they have a great impact on the child's psychological and emotional development.

However, every parent seeks for a rapid and easy treatment for their children, but if the child is uncooperative that will require multiple dental visits , more expenses or he/she might undergo general anesthesia which is more expensive.

Also, the parent-child relationship is very important ,bad relationship can cause insecurities, lack of self confidence and trust, resulting in the future a fearful and irresponsible man / woman.

ELIGIBILITY:
Inclusion Criteria:

* children with Primary teeth
* Before the eruption of permanent molar
* First dental visit
* Both genders

Exclusion Criteria:

* Children with systemic diseases or congenital problems
* Parents refuse to participate

Ages: 3 Years to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children with primary dentition during their first dental visit and their parents or caregiver
Sampling Method: Probability Sample
Enrollment: 1 (Estimated)
Dates: Start 2020-05 (Estimated); Primary Completion 2021-06 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Parenting style | 1 year
  There are four types of parenting styles :authoritative, authoritarian, permissive and neglecting. Each parent or caregiver will be asked to fill a questionnaire which includes multiple behavior and actions exhibited by the parents and they will do rating for each item how often they exhibit this behavior and accordingly will determine which parenting style they belong to.
  There are five scales or ratings :
  1. Never
  2. Once in a While
  3. About Half the Time
  4. Very Often
  5. Always

SECONDARY OUTCOMES:
Behavior of children | 1 year
  Behavior of children will be videotaped and monitored according to Frankl scale.
  Frankl scale is a way to assess the child's behavior during his dental visits.There are four scales either definitely negative, or negative, or positive, or definitely positive.
  1. -/- Definitely Negative. Refusal of treatment, forceful crying, fearfulness, or any other evidence of extreme negatism.
  2. - Negative. Reluctance to accept treatment, uncooperative, some evidence of negative attitude but not pronounced (sullen, withdrawn).
  3. + Positive. Acceptance of treatment; cautious behavior at times; willingness to comply with the dentist, at times with reservation, but patient follows the dentist's directions cooperatively
  4. +/+ Definitely positive. Good rapport with the dentist, interest in the dental procedures, laughter and enjoyment.

REFERENCES:
- [Background] Howenstein J, Kumar A, Casamassimo PS, McTigue D, Coury D, Yin H. Correlating parenting styles with child behavior and caries. Pediatr Dent. 2015 Jan-Feb;37(1):59-64. PMID 25685975
- [Background] Park H, Walton-Moss B. Parenting style, parenting stress, and children's health-related behaviors. J Dev Behav Pediatr. 2012 Jul;33(6):495-503. doi: 10.1097/DBP.0b013e318258bdb8. PMID 22772823
- [Background] Aminabadi NA, Farahani RM. Correlation of parenting style and pediatric behavior guidance strategies in the dental setting: preliminary findings. Acta Odontol Scand. 2008 Apr;66(2):99-104. doi: 10.1080/00016350802001322. PMID 18446551